CLINICAL TRIAL: NCT01859650
Title: Lung HeXeRT: Advanced Proton, Hyperpolarised 3-helium and 129-xenon Magnetic Resonance Imaging for Lung Cancer Radiotherapy Planning and Evaluation
Brief Title: Lung HeXeRT: Helium, Xenon MRI for NSCLC Patients
Acronym: HeXeRT
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); Weston Park Hospital Cancer Charity (Other); Sheffield Hospitals Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: STH17245
Record Dates: First submitted 2013-05-10; First posted 2013-05-22 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NSCLC patients undergoing RT
  Interventions: Other: MR and CT imaging

INTERVENTIONS:
Other: MR and CT imaging

SUMMARY:
The University of Sheffield is one of the leading centres in the world for basic and translational research with inhaled gas MRI, which provides lung images with unprecedented spatial and temporal resolution. Our previous work demonstrated that inhaled gas MRI can provide significant clinical information for lung cancer radiotherapy planning and post-treatment evaluation. Building upon this unique experience, a multidisciplinary team will conduct an inhaled gas and proton lung MRI study that will address two of the major clinical problems faced by lung cancer patients treated with radiotherapy.

1. Normal lung tissue is often damaged by the curative radiation dose. The investigators hypothesise that regional ventilation-perfusion lung function imaging with inhaled gas and proton MRI before and after treatment will help to lower the risk of radiation-induced lung injury and help to detect such damage at an early stage.
2. Identification of the extent of cancerous tissue is error-prone when planning treatment from CT images alone. The investigators hypothesise that advanced proton MRI techniques will improve the identification of tumour volume, which is critical to successfully targeting the radiation dose.

To achieve these goals, image acquisition and image processing methods will be tested with a study of 20 patients. Results from this study will make an important contribution to improving the treatment of lung disease which is one of the key research priorities of the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an MDT diagnosis of NSCLC based on findings of positive histology, positive PET scan or growth on serial CT scan requiring CT planning for radiotherapy treatment
* patients aged over 18
* patients able to undergo MRI scanning.

Exclusion Criteria:

* patients with co-morbid conditions that exclude radiotherapy treatment
* patients who are pregnant or women with child bearing potential
* patients unable to give informed consent
* patients who do not understand English sufficiently to read the patient information sheet, provide informed consent or converse with research staff without interpreters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC attending Weston Park Hospital, Sheffield, UK.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of ventilated lung measured using inhaled gas MRI | Change between pre treatment (average 10 days before start of treatment) and at 3 months post treatment

SECONDARY OUTCOMES:
Lung tumour volume measured using proton MRI | Change between pre-treatment (average 10 days before start of treatment) and at 3 months post treatment
Percentage of ventilated lung measured using CT | Change between pre-treatment (average of 10 days before start of treatment) and at 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Q Hatton, FRCR, FRCP, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

REFERENCES:
- [Background] Wild JM, Ajraoui S, Deppe MH, Parnell SR, Marshall H, Parra-Robles J, Ireland RH. Synchronous acquisition of hyperpolarised 3He and 1H MR images of the lungs - maximising mutual anatomical and functional information. NMR Biomed. 2011 Feb;24(2):130-4. doi: 10.1002/nbm.1565. Epub 2010 Sep 6. PMID 20821726
- [Background] Ireland RH, Din OS, Swinscoe JA, Woodhouse N, van Beek EJ, Wild JM, Hatton MQ. Detection of radiation-induced lung injury in non-small cell lung cancer patients using hyperpolarized helium-3 magnetic resonance imaging. Radiother Oncol. 2010 Nov;97(2):244-8. doi: 10.1016/j.radonc.2010.07.013. Epub 2010 Aug 17. PMID 20724011
- [Background] Bates EL, Bragg CM, Wild JM, Hatton MQ, Ireland RH. Functional image-based radiotherapy planning for non-small cell lung cancer: A simulation study. Radiother Oncol. 2009 Oct;93(1):32-6. doi: 10.1016/j.radonc.2009.05.018. Epub 2009 Jun 22. PMID 19552978
- [Background] Ireland RH, Woodhouse N, Hoggard N, Swinscoe JA, Foran BH, Hatton MQ, Wild JM. An image acquisition and registration strategy for the fusion of hyperpolarized helium-3 MRI and x-ray CT images of the lung. Phys Med Biol. 2008 Nov 7;53(21):6055-63. doi: 10.1088/0031-9155/53/21/011. Epub 2008 Oct 9. PMID 18843168
- [Background] Ireland RH, Bragg CM, McJury M, Woodhouse N, Fichele S, van Beek EJ, Wild JM, Hatton MQ. Feasibility of image registration and intensity-modulated radiotherapy planning with hyperpolarized helium-3 magnetic resonance imaging for non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):273-81. doi: 10.1016/j.ijrobp.2006.12.068. PMID 17448880